CLINICAL TRIAL: NCT04836598
Title: Bikini Scarless Laparoscopic Cholecystectomy for Morbid Obesity as a Day Case.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Bassem Mohamed Sieda, assistant professor of general surgeryt, Zagazig University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 11671
Record Dates: First submitted 2021-03-31; First posted 2021-04-08 (Actual); Last update posted 2021-04-08 (Actual); Status verified 2021-04

CONDITIONS: Cholecystitis, Chronic
Keywords: scarless cholecystectomy; Breif port cholecystectomy
MeSH Terms: conditions — Cholecystitis; Bronchiolitis Obliterans Syndrome | interventions — Cholecystectomy, Laparoscopic

STUDY DESIGN:
Intervention Model Description: Patients were randomly allocated into 2 groups (Consort Chart) and each group categorized into 3 subgroups according to BMI, into class I: Obese Class 1 30-34.9kg/m2, Class II: Obese Class II 35-39.9kg/m2 and class III: Morbidly Obese Class III >40kg/m2
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Multiport laparoscopic cholecystectomy (Active Comparator): controlled group
  Interventions: Other: laparoscopic cholecystectomy
- Bikini line laparoscopic cholecystectomy (Active Comparator): bikini line 2 ports
  Interventions: Other: laparoscopic cholecystectomy

INTERVENTIONS:
Other: laparoscopic cholecystectomy — A Prospective randomized controlled trial study was undertaken along 4 years Between November 2016 and October 2020, in two institutions. 400 patients were selected, 200 patients underwent BLLC and 200 patients underwent multiple port laparoscopic cholecystectomy (MPLC).
  Other Names: brief port scarless laparoscopic cholecystectomy

SUMMARY:
Background: Bikini line laparoscopic cholecystectomy is a safe method, used as a scarless cosmetic port technique for gall bladder diseases in morbid obese patients as a day case.

Objectives:

The aim of this study was to investigate the safety and efficacy of an elective Bikini line laparoscopic cholecystectomy in the morbid obese patients with chronic calcular cholecystitis, and review our experience with Bikini line laparoscopic cholecystectomy as minimal invasive scarless technique.

We issued a modifications in order to minimize the number of ports (Brief ports) and modify port sites, using the Bikini line laparoscopic cholecystectomy as a cosmetic and hidden scar laparoscopy for obese patients concerned with aesthetic results and body image. Aiming at faster recovery, decrease pain and improve cosmoses.

Bikini Line laparoscopic cholecystectomy is technically safe and effective day surgery procedure for chronic cholecystitis patients with higher patient satisfaction regarding pain and cosmoses. Obesity, intended as BMI 40, does not have any obstacle on the technical feasibility of BLLC.

DETAILED DESCRIPTION:
Thoroughly, BLLC is a novel technique aimed at solving the issue of cosmoses that is always presented as a main complaint from morbid obese patients. The main concern to use Brief ports laparoscopy or hidden scar laparoscopy to reduce incisions and change sites. The study designed to identify superiority of technique regarding success as a day case surgery, better cosmoses and lesser pain.

We tried to wear off the port sites scar and kept our stabs in the suprapubic Bikin line. We kept camera port in the navel's natural scar and used the other ports in lower abdominal crease at Bikini line. Cosmosis has been and still the reason among patient population to accept the laparoscopic surgery, many synonyms can be applied here, as Cosmotic,Hidden scar, Scarless, Non-visualized or Scarless Bikini cholecystectomy.

BLLC is performed under general anesthesia. Patient placed in the supine position with patient's legs apart and arms are rolled in, patient strapped to table at the mid-thigh. Surgeon stood between patient's legs, the camera man stood on the right side of patient, monitor placed near patient head to the right side. Three ports were used, 12 mm visiport (….) umbilical, with A 30 degree camera used, 5mm in Bikini line at Right mid-clavicular line and third port 5mm in Bikini line at left mid-clavicular line (Figure) Patient kept in reverse Trendlenburg position with maximum degree 20. But to lesser degree than done in classic LC,

ELIGIBILITY:
Inclusion Criteria:

* Morbid obese patients with BMI ≤30 KG/M2 and ≥ 40 9kg/m2 with symptomatic uncomplicated gall stones, ASA 1-3.

Exclusion Criteria:

* Acute calcular cholecystitis, BMI ≥45, ASA 4 or higher, length of stay more than 1 day.

Patients required additional trocars for patient safety, readmission,

Ages: 17 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 3 (Estimated)
Dates: Start 2016-11-30 (Actual); Primary Completion 2021-04-20 (Estimated); Study Completion 2021-04-30 (Estimated)

PRIMARY OUTCOMES:
a successful and safe day case | 4 years
  a successful and safe day case laparoscopic cholecystectomy with discharge on the same day with no significant pain.
  patient stayed more than a day was not enrolled

SECONDARY OUTCOMES:
Measured patient satisfaction from body image and cosmoses within 6 months from surgery. | 3 years
  Postoperative pain was defined as mild, moderate sever according to visual analogue scale (VAS)
  Pain assessment at the tommy and at port sites were assessed at postoperative day 1 and at discharge as follow, 8 hours, at discharge time at 12 hours or 24 hours postoperative, and after discharge at 48 hours, 72 hours achieved through Telephone call with the patient.
  Patient satisfaction from cosmetic outcome was measured on 10 points scale. Divided into mild satisfied (1-3 points), moderate (4-7)and highly satisfied (8-10 points) at the second postoperative visit at 30 days postoperative, after 3 months and after 6 months, based on patient question to rate it, mild satisfaction: 1-3, moderate satisfaction:4-7 and highly satisfied: from 8-10

CONTACTS AND LOCATIONS:
Overall Officials: Bassem M Sieda, professor, Study Chair — 1975
Locations (3):
- Zagazig University hospitals, Zagazig, Outside USA, Egypt
- Saudi Arabia (2):
  - Saudi German hospital, Riyadh, Outside USA
  - Saudi german hospital, Riyadh

IPD SHARING:
Plan to Share IPD: Yes
data can be shared through the publisher and all authers
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 1 year
Access Criteria: publisher which is international journa